CLINICAL TRIAL: NCT01073800
Title: Using AtorVASTatin to Prevent VAscular Inflammatory OccLUSion in the Critically Ill
Acronym: VASTVALUS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VASTVALUS
Record Dates: First submitted 2009-07-20; First posted 2010-02-23 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Myocardial Infarction; Stroke; Renal Failure
Keywords: atorvastatin; vascular occlusion; myocardial infarction; stroke; renal failure; critically ill; Vascular occlusive events among the critically ill
MeSH Terms: conditions — Myocardial Infarction; Stroke; Renal Insufficiency; Critical Illness | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atorvastatin 80 mg (Active Comparator): active treatment
  Interventions: Drug: atorvastatin 80 mg per os daily
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atorvastatin 80 mg per os daily — atorvastatin 80 mg per os daily
  Arms: atorvastatin 80 mg
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
Patients are admitted to the critical care unit of the hospital because of medical conditions that have a high likelihood of causing severe problems with blood flow, breathing, or brain function. These conditions also have a high likelihood of causing death. Approximately 10 to 15% of all critically ill patients die in hospital. A large amount of scientific evidence suggests that a substantial proportion of these deaths is due to a combination of blot clotting and inflammation in the blood vessels.

Statins are drugs that interfere with cholesterol and fat metabolism. Cholesterol and fat in the blood are associated with blood clotting and inflammation in the blood vessels. Statins are known to be very beneficial in improving the survival after heart attacks, and in preventing heart attacks.

The question that VASTVALUS asks is: do statins improve survival among all critically ill patients? In VASTVALUS, we will concentrate on patients that do not currently require a statin because of their medical condition e.g. after a heart attack, but we are concerned with the rest of the critically ill. In VASTVALUS, participating patients will receive either atorvastatin 80 mg daily or a placebo. Atorvastatin is a statin with a well-established record of safety and effectiveness. A placebo has no known medical activity. We will follow all patients in VASTVALUS to determine whether atorvastatin has any effect on the occurrence of death, stroke, heart attack, or kidney failure among the critically ill. Results from VASTVALUS will be shared with the medical community after the study is completed. As with all clinical trials, patients in VASTVALUS participate of their own choice, and can change their mind at any time.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men or women >18 years of age
* 2. Admitted to a critical care unit and requiring at least a 48 hour critical care unit stay for medical reasons. Medical reasons include:

  * conditions of cardiovascular,
  * respiratory, or
  * neurologic impairment that require supportive care and observation.

Exclusion Criteria:

* 1. Hepatic failure (Childs-Pugh class C)
* 2. Rhabdomyolysis
* 3. Allergy or hypersensitivity to this drug or any of its components
* 4. Previous intolerance
* 5. Enrolment in another interventional trial
* 6. Contraindication to gastric and/or small bowel drug administration
* 7. MI as major diagnosis at admission (statin indicated)
* 8. Coronary artery intervention within previous 3 days
* 9. Currently receiving a statin or indicated (MI, dyslipidemia)
* 10. Pregnancy
* 11. personal or family history of hereditary muscular disorders
* 12. previous history of muscle toxicity with another HMG-CoA reductase Inhibitor
* 13. concomitant use of a fibrate or niacin
* 14. hypothyroidism
* 15. alcohol abuse
* 16. excessive physical exercise
* 17. renal impairment
* 18. diabetes with hepatic fatty change
* 19. surgery and trauma
* 20. frailty
* 21. situations where an increased plasma level of active ingredient may occur

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
vascular occlusive events | 30 days

SECONDARY OUTCOMES:
liver enzyme elevation | 30 days
rhabdomyolysis | 30 days
myalgias | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada